CLINICAL TRIAL: NCT05473754
Title: Feasibility Study About Super Digital Platform: a Joint System for Rehabilitation and Educational Projects for Children With Autism Spectrum Disorder
Brief Title: Super: a Joint System in a Rehabilitation Educational Digital Platform
Acronym: SUPER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Giulia Purpura, PhD, Researcher, University of Milano Bicocca
Other Study IDs: SUPER
Record Dates: First submitted 2022-05-09; First posted 2022-07-26 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Autism Spectrum Disorder; Telerehabilitation
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: Families, teachers, and clinicians use SUPER digital platform in addition to usual rehabilitative and educative interventions.
  Interventions: Behavioral: SUPER digital platform
- Control Group: Families, teachers, and clinicians perform usual rehabilitative and educative interventions.

INTERVENTIONS:
Behavioral: SUPER digital platform — SUPER digital platform was implemented to ensure synergy between ASD families, health services, and schools through different tools to share rehabilitative and educational objectives and strategies. It was designed following the ASD International Guidelines and the recommendations of the ICF-CY and was organized into two areas: General (to promote scientific knowledge on ASD) and Personalized (restricted virtual space for groups of users following an individual with ASD).
  Groups: Experimental Group

SUMMARY:
Due to its complexity and variability, Autism Spectrum Disorder (ASD) requires multidisciplinary and multidimensional interventions. SUPER (in Italian: Sistema Unitario in una Piattaforma Riabilitativa ed Educativa) is an Italian digital platform, implemented to facilitate collaboration between families, health services, and schools and to promote personalized intervention for children with ASD. The research protocol, aimed to test SUPER's feasibility and usability, foresees the enrollment of 12 ASD children in the Experimental Group (EG) and 12 ASD children for the Control Group. All families, teachers, and clinicians will perform usual rehabilitative and educative interventions, but the EG will use SUPER, in addition to ordinary programs. The feasibility and acceptability of SUPER will be assessed through usability scales and questionnaires realized ad hoc for the purpose. At baseline and established endpoints, ASD patients will be evaluated with different assessment tools.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder
* Access to Child Neuropsychiatry or Pediatric Rehabilitation services participating in the study
* Age of patients from 3 to 7,11 years
* Informed consent freely acquired before the start of the study by the patient's parents

Exclusion Criteria:

* Patients with severe genetic degenerative diseases
* Patients with severe sensory disabilities
* Patients with severe medical complications

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Autism Spectrum Disorders that perform rehabilitative programs
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-09-09 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline at 3 months in a specific questionnaire that evaluates perception of taking charge | T0 (baseline) and T1 (after 3 months)
  Questionnaire created ad hoc for taking charge: it is a parent-report instrument with 22 items based on a 5-points Likert Scale. Higher scores (maximum 110) mean a better perception of taking charge, while lower scores (minimum 22) mean a worse perception about taking charge.
Acceptability of SUPER Digital Platform | T1 (after 3 months of use of SUPER by parents, clinicians and teachers)
  SUPER Questionnaire is an instrument created ad hoc to evaluate the acceptability of SUPER platform for parents, clinicians and teachers of children with ASD. It is composed by 38 items based on a 5-points Likert Scale. Higher scores (maximum 190) mean optimal acceptability of SUPER within the rehabilitative taking charge, while lower scores (minimum 38) mean a worse level of acceptability.
Usability of SUPER Digital Platform via System Usability Scale | T1 (after 3 months of use of SUPER by parents, clinicians and teachers)
  SUS (System Usability Scale) is a standardized tool for measuring the perceived usability of an interactive system, such as websites, user interfaces, and web applications. It consists of 10 items that are scored on a Likert scale, from 1 (strongly disagree) to 5 (strongly agree). The SUS scores below 68 reveal usability issues with the system, while scores higher than 68 indicate acceptable levels of usability. More specifically, scores over 80 suggest an "excellent" usable system, scores between 68 and 80 can be considered "good", scores between 51 and 68 indicate "fair" results, scores below 51 are "poor", and scores below 36 reflect "unusable" systems.
Change from baseline at 3 months in the Parent Stress Index-Short Form (PSI-SF) | T0 (baseline) and T1 (after 3 months)
  The Parenting Stress Index-Short Form (PSI-SF) is one of the most commonly used measures of parenting stress both in clinical and research contexts. The PSI-SF is a 36-item, self-report measure with three subscales: Parental Distress (PD), Parent-Child Dysfunctional Interaction (PCDI), and Difficult Child (DC). Items are scored using the following 5-point scale: 1) SA (Strongly Agree); 2) A (Agree); 3) NS (Not Sure); 4) D (Disagree); 5) SD (Strongly Disagree).The normal range of scores is between the 15th and 80th percentile. Scores at or above the 85th percentile are considered high and Defensive Reponding scores at 10 or below are considered extremely low.

SECONDARY OUTCOMES:
Efficacy of SUPER Digital Platform to support rehabilitation about adaptive behaviour in children with ASD by VABS-2 | T0 (baseline), T2 (after 6 months)
  Vineland Adaptive Behavior Scales- 2 (VABS-2) is designed to measure adaptive behavior in daily settings for children and adults from birth to 90 years of age. The Vineland-II items are arranged from 11 simple to more complex behavior subdomains across four main domains: Communication, Daily Living Skills, Socialization, and Motor Skills. It also provides an optional Maladaptive Behavior Index. Items are arranged in a developmental sequence within each subdomain, with each item rated on a 3-point scale (i.e., 0 = Behavior Never Performed, 1 = Behavior Sometimes or Partially Performed, or 2 = Behavior Usually or Habitually Performed).
  The Adaptive Behavior Composite and domains yield age-based standard scores with a normative M=100 and SD=15, and subdomains yield standard scores with a M=15 and SD=3.
Efficacy of SUPER Digital Platform to support rehabilitation about behaviour of ASD children by CBCL | T0 (baseline), T1 (after 3 months); T2 (after 6 months)
  Child Behavior Checklist (CBCL) is a standardized questionnaires that provides information on six scales: affective problems, attention-deficit/hyperactivity, anxiety, oppositional defiance, somatic problems, and conduct problems. It has two separate forms, one for children 1.5-5 years old and one for children 6-18 years old. On both versions, there is a Total Problems score, as well as composites for Internalizing and Externalizing Problems. DSM-Oriented Scales were formed based on experts' ratings of how well the items fit DSM criteria for relevant Major and Dysthymia for Affective Problems, Anxiety Problems, Oppositional Defiant Problems, and Conduct Problems. The preschool version the DSM-Oriented scales are for Affective Problems, Anxiety Problems, Pervasive Developmental Problems, Attention-Deficit/Hyperactivity Problems, and Oppositional Defiant Problems.
Efficacy of SUPER Digital Platform to support the improvement of autistic symptoms in ASD children by CARS-2 | T0 (baseline), T2 (after 6 months)
  Childhood Autism Rating Scale - Second Edition (CARS-2) is extremely useful in identifying symptoms of autism. The clinician rates the individual on each item (15 items), using a 4-point response scale. Ratings are based not only on the frequency of the behavior in question, but also on its intensity, peculiarity, and duration.Scores above the cutoff (28) can be broken down into "mild-to-moderate" level of autistic behaviors vs. "severe" level.
Efficacy of SUPER Digital Platform to support the improvement of social communication ASD children by SCQ | T0 (baseline), T1 (after 3 months), T2 (after 6 months)
  SCQ is a parent-report tool to evaluate communication skills and social functioning in children who may have autism or autism spectrum disorders. The questionnaire is composed of just 40 yes-or-no questions. Both forms can be given directly to the parent, who can answer the questions without supervision. Higher scores mean a worse functioning. It produces results that can be helpful in treatment planning, educational intervention, and measurement of change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Renata Nacinovich, MD, Principal Investigator — University of Milano Bicocca
Locations (2):
- Italy (2):
  - ASST Monza, University of Milano Bicocca, Monza
  - Centro Riabilitativo Pompei, Pompei

IPD SHARING:
Plan to Share IPD: Undecided